CLINICAL TRIAL: NCT03925636
Title: Treatment With the Specific Carbohydrate Diet for Children With Clostridium Difficile Colonization
Brief Title: Specific Carbohydrate Diet for Clostridium Difficile
Acronym: SCD_cDiff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Suskind (Other)
Collaborators: Pacific Northwest National Laboratory (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Suskind, Professor of Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15858
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Clostridium Difficile Infection; Diet Modification
Keywords: Specific Carbohydrate Diet; Clostridium Difficile Infection; Clostridium Difficile; cDiff; Diet
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary therapy for C. difficile colonization (Experimental): Dietary therapy intervention for this arm is the Specific Carbohydrate Diet.
  Interventions: Dietary Supplement: Specific Carbohydrate Diet

INTERVENTIONS:
Dietary Supplement: Specific Carbohydrate Diet — The diet removes all grains such as wheat, barley, corn, rice, and most dairy products (except yogurt fermented for 24 hours and cheese aged for grater than 30 days). The diet mainly consists of meat, fruits, vegetables, nuts, oils, and honey.

SUMMARY:
The investigators are doing this research study to answer questions about a nutritional therapy called the Specific Carbohydrate Diet (SCD) for children with active Clostridium Difficile Infection.

For this study, the investigators will be looking to determine:

1. Is SCD effective for the treatment for Clostridium Difficile Colonization?
2. Is the SCD well tolerated?

DETAILED DESCRIPTION:
The aim of this study is to determine the tolerability and potential efficacy of dietary therapy, the Specific Carbohydrate Diet (SCD), in pediatric patients with persistent antigen positivity due to C. difficile colonization with minimally active symptomatology. The goal of this pilot study is to gather preliminary data for a future treatment controlled trial of SCD versus standard medical therapy.

This is a single center, open labelled study designed to determine tolerability, preliminary safety and potential efficacy in pediatric patients with persistent C. difficile colonization with minimally active symptomatology. The study patients will be recruited from Seattle Children's Gastroenterology and Infectious Disease clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents eighteen months old to twenty one years old
2. Diagnosis of C. difficile based upon stool antigen and toxin
3. Minimally active symptomatology based upon

   1. 4 or less stools per day
   2. No evidence of dehydration
   3. No evidence of bandemia or hypoalbuminemia on screening labs
4. Parent/guardian and child must be able to comprehend the consent and assent
5. Parent/guardian and participant must be able to attend study visits at baseline, and weeks +2, +4, +8, +12.
6. Patient must not have had antibiotic treatment directed at C. difficile for at least 1 week.

Exclusion Criteria:

1. Severe symptoms

   1. Abdominal pain that interrupts or inhibits normal activity
   2. Fever
   3. Vomiting
   4. Blood in stool
2. Clinical signs of coexisting acute systemic illnesses (meningitis, sepsis, pneumonia), immunodeficiency, underlying severe chronic diseases, and cystic fibrosis
3. Tobacco, alcohol or illicit drug abuse
4. Currently taking antibiotics at time of enrollment
5. Malnutrition as judged by the ratio of weight to height,
6. Clinical signs of dehydration(CD score>0)

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with negative C. difficile stool | 12 weeks
  Stool is analyzed for C. difficile antigen and toxin by enzyme-linked immunosorbent assay (EIA). Samples that are antigen positive and toxin negative by EIA screen will be analyzed by the more sensitive polymerase chain reaction amplification (PCR) assay to detect C. difficile toxin.
Number of participants able to maintain the specific carbohydrate diet | 4 weeks
  Diet diaries are reviewed to ascertain compliance to diet. Questionnaires are reviewed to determine barriers to implementing the diet.

CONTACTS AND LOCATIONS:
Overall Officials: David L Suskind, MD, Principal Investigator — Seattle Children's Hospital and The University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Not discussed

REFERENCES:
- [Background] Suskind DL, Wahbeh G, Gregory N, Vendettuoli H, Christie D. Nutritional therapy in pediatric Crohn disease: the specific carbohydrate diet. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):87-91. doi: 10.1097/MPG.0000000000000103. PMID 24048168
- [Background] Suskind DL, Lee D, Solan P, Wahbeh G, Hayden H, Brittnacher M, Nuding M, Miller S. Dietary therapy for clostridium difficile colonization: A case series. Anaerobe. 2019 Jun;57:1-3. doi: 10.1016/j.anaerobe.2019.02.016. Epub 2019 Feb 28. PMID 30826445
- See also: Case Series of dietary therapy for recurrent c. difficile and colonization — https://www.ncbi.nlm.nih.gov/pubmed/30826445

DOCUMENTS (1):
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03925636/ICF_000.pdf